CLINICAL TRIAL: NCT06882707
Title: The Effectiveness of Neurodynamic Nerve Mobilization in Addition to Physical Therapy on the Median Nerve and Abductor Pollicis Brevis Muscle in Patients With Mild and Moderate Carpal Tunnel Syndrome
Brief Title: The Effectiveness of Neurodynamic Mobilization in Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Merve Akdeniz Leblebicier, MD, Kutahya Health Sciences University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: MedianNerveMobilization
Record Dates: First submitted 2025-03-12; First posted 2025-03-18 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Carpal Tunnel Syndrome (CTS); Median Nerve
Keywords: carpal tunnel syndrome; median nerve mobilization; abductor pollicis brevis; boston carpal tunnel questionnaire; hand grip; ultrasonography
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Ultrasonic Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Median nerve mobilization in addition to ultrasound therapy (Experimental): In addition nerve mobilization, ultrasound therapy will be applied to all patient in experimental group via methods explained below.
  Interventions: Other: Median Nerve Mobilization; Other: Ultrasound therapy
- Ultrasound therapy (Active Comparator): In control group, patients will received only ultrasound therapy.
  Interventions: Other: Ultrasound therapy

INTERVENTIONS:
Other: Median Nerve Mobilization — Passive neuromobilisation of the median nerve and functional self-exercises. The procedure started with the patient in the supine position. The following steps were taken in sequence: shoulder girdle depression; slight abduction of the elbow extension with arm lateral rotation and forearm supination; wrist, finger and thumb extensions were added; and the shoulder was taken into further extension.
  To apply maximum stretch opposite cervical side flexion was done, and, in the end, the wrist was repeatedly moved into and out of stretch by performing a few degrees of flexion and extension at the wrist.
  This mobilization technique will be performed by an experienced physician/physiotherapist three times a week for 3 weeks, and the patients will be given 3 sets of 15 cycles with a 1-minute rest period in each set.
  Arms: Median nerve mobilization in addition to ultrasound therapy
Other: Ultrasound therapy — In control group, patients will received only ultrasound therapy. The patient will be in a sitting position with his/her face facing the physiotherapy technician, elbow in 90 degree flexion, forearm in supination, wrist in neutral position and supported by placing a towel under the patient's extremity and will be applied in Us intermittent mode with an intensity of 0.8 W/cm2 in 1 MHZ frequency in 1:4 mode for 10 minutes, moving in a way to draw an infinity sign for 10 seconds. Treatment will be given 5 days a week for 3 weeks and a total of 15 sessions.

SUMMARY:
This randomized, clinical, single-blinded, controlled study will initially planned to include 86 patients diagnosed with carpal tunnel syndrome who applied to Kütahya Health Sciences University, Evliya Çelebi Training and Research Hospital, Physical Medicine and Rehabilitation outpatient clinic and Kutahya City Hospital.Patients aged 20-55 years who were diagnosed with mild and moderate carpal tunnel syndrome by electromyography (EMG) in the last 6 months were included in the study. The patients were randomized into two groups using the computer-assisted randomization method. Median nerve mobilization and ultrasound therapy will be given to the study group, and only ultrasound therapy will be given to the control group. All the patients were evaluated with the Visual Analog Scale (VAS), Hand and Pinching Grip Test, Boston Carpal Tunnel Questionnaire (BCTQ) and Median Nerve and Abductor Pollicis Brevis Muscle ultrasonography before the intervention and at the third week of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with mild-to-moderate CTS on the dominant hand, based on the electrodiagnostic examination.
* Aged 20-55 years.
* Consent to receive the described treatment.
* Lasting symptoms at least 3 months

Exclusion Criteria:

* A systemic inflammatory disease.
* Any disease that can cause polyneuropathy, for example, diabetes mellitus.
* A cognitive disorder.
* Receiving psychotherapy.
* A pacemaker.
* Any disease that can affect the central nervous system.
* Carpal tunnel syndrome surgery history

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2025-03-15 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Ultrasound assessment | Change from Baseline at 3th weeks
  The Median nerve's diameter will be evaluated bilaterally by another researcher blinded to interventions and experienced in musculoskeletal ultrasonography, using ultrasound with a 6-18 Mhz linear probe (Mindray-UMT 200, USA).
  During the examination, patients will be seated on a stretcher, while the examiner sat on a higher stool.
  The Median nerve will be evaluated by measuring the circumference of the nerve at the location where the nerve entered the carpal tunnel.
  The ultrasound probe will be positioned above the epicondylus lateralis. The nerve cross-sectional area (CSA) will be recorded in the carpal tunnel while it was perpendicular to the wrist at 90 degrees on the Median nerve trace.
  The nerve diameter will be measured from the circumference of the epineurium.

SECONDARY OUTCOMES:
Hand and pinching grip measurement | Change from Baseline at 3th weeks
  The grip strength of the hand is measured with the Jamar hand dynamometer recommended by the American Association of Hand Therapists (AETD).
  The measurement will be performed in the standard position specified by the AETD; the patient will be seated, shoulders in adduction and neutral rotation, elbow in 90 degree flexion, forearm in mid-rotation and supported, wrist in neutral position with three repetitions and the results will be recorded in kilograms.
  Pinch force will be measured in the same position as the hand grip strength is measured with a pincmeter.
  It will be evaluated in two different positions, lateral and triple grip. When evaluating the lateral grip, the patient will be asked to press the pinchmeter from the top with the middle of the distal phalanx of the thumb and support the lower part of the pinchmeter with the second phalanx of the index finger.
  When evaluating the triple grip, measurements will be made by squeezing the thumb on one side of the pinchmeter an
Symptom severity and functional status | Change from Baseline at 3th weeks
  Symptom severity and functional status were evaluated with BCTQ, a self-report measure of CTS with two domains: the Boston Carpal Tunnel Syndrome Questionnaire Symptom severity scale comprising 11 items to evaluate pain, paresthesia, and weakness and the Boston Carpal Tunnel Syndrome Questionnaire Symptom functional status domain with eight items assessing the ability to perform hand-related activities.
  For each item, a high score indicates an increasing severity of symptoms or difficulty experienced.
  The validity and reliability analyses of the Turkish version of BCTQ were undertaken by Sezgin et al19 Reliability of the Turkish version was very good, with high internal consistency (Cronbach's alpha 0.82 for symptom severity scale, and 0.88 for functional status scale), and reproducibility (Pearson correlation coefficient 0.60 for symptom severity scale, and 0.77 for functional status scale).

CONTACTS AND LOCATIONS:
Overall Officials: Merve Akdeniz LEBLEBİCİER, MD, Principal Investigator — Kutahya Health Sciences University
Locations (1):
- Kutahya Health Sciences University, Kütahya, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No